CLINICAL TRIAL: NCT04235751
Title: Effect of Coaching on Surgeon Well-Being, Job Satisfaction, & Fulfillment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Liselotte (Lotte) N. Dyrbye, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19-011708
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Professional Burnout; Professional Stress; Job Stress
MeSH Terms: conditions — Burnout, Professional; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Coaching Intervention (Experimental): Subjects will receive 6 professional coaching sessions
  Interventions: Behavioral: Professional Coaching
- Delayed Coaching Intervention (Experimental): Subjects will receive no coaching for the first six months of the study, at which point they cross over and receive 6 professional coaching sessions
  Interventions: Behavioral: Professional Coaching

INTERVENTIONS:
Behavioral: Professional Coaching — 6 individualized professional coaching sessions via phone

SUMMARY:
Researchers are trying to determine if individualized professional coaching improves physicians' sense of well-being and job satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons at Mayo Clinic

Exclusion Criteria:

* Retired surgeons at Mayo Clinic; physicians in other disciplines or organizations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Burnout | Baseline, 6 months
  Change in self-reported Maslach Burnout Inventory (MBI) Score using a scale of never, a few times a year or less, once a month or less, a few times a month, once a week, a few times a week, every day
Job Satisfaction | Baseline, 6 months
  Change in self-reported Physician Job Satisfaction Scale score using a scale of 1=very strongly disagree to 5= very strongly agree
Professional Fulfillment | Baseline, 6 months
  Change in the self-reported Empowerment at Work Scale score using a scale of 1=very strongly disagree to 7=very strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte N Dyrbye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dyrbye LN, Gill PR, Satele DV, West CP. Professional Coaching and Surgeon Well-being: A Randomized Controlled Trial. Ann Surg. 2023 Apr 1;277(4):565-571. doi: 10.1097/SLA.0000000000005678. Epub 2022 Aug 24. PMID 36000783
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials